CLINICAL TRIAL: NCT03510598
Title: Fat Reduction in the Submental Area - a Sequential Treatment Approach With CoolMini and KYBELLA®
Brief Title: Submental Study (Sequential Treatment Approach)
Acronym: CMK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZA17-005
Record Dates: First submitted 2018-04-10; First posted 2018-04-27 (Actual); Results first posted 2021-12-30 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2020-08

CONDITIONS: Body Fat Disorder
MeSH Terms: interventions — Deoxycholic Acid; Injections

STUDY DESIGN:
Intervention Model Description: Kybella and Zeltiq CoolSculpting CoolMini
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment for Submental Fat Reduction withCoolSculpting System followed by Kybella (Experimental): CoolSculpting followed by Kybella treatments. Kybella supplied in 2mL vials.
  Interventions: Device: The ZELTIQ CoolSculpting System; Drug: Kybella 20 MG in 2 ML Injection

INTERVENTIONS:
Device: The ZELTIQ CoolSculpting System — The CoolSculpting machine will be used to perform the treatments.
Drug: Kybella 20 MG in 2 ML Injection — Injectable drug called KYBELLA® (deoxycholic acid)

SUMMARY:
Evaluate the safety and efficacy of subcutaneous fat layer reduction in the submental area using multiple therapeutic tools.

DETAILED DESCRIPTION:
The Zeltiq CoolSculpting System and the sequential use of the injectable drug Kybella for non-invasive and then minimally invasive fat reduction in the submental area will be evaluated during the study.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects > 22 years of age and < 65 years of age.
* Women of childbearing potential must have a negative urine pregnancy test result at screening and agree to practice adequate contraception.
* CR-SMFRS grade of 4 (extreme) as determined by the evaluating investigator at screening.
* Dissatisfaction with the submental area expressed by the subject as a rating of 0, 1 or 2 using the Subject Self Rating Scale (SSRS) as determined at Screening visit.
* History of stable body weight confirmed by the subject, for at least 6 months prior to the first treatment session.
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the course of the study.
* Subject agrees to forgo any treatment or behavior (e.g., unshaven facial hair) during the subject's participation in the study that may affect the assessments of the submental area.
* Subject is medically able to undergo the administration of KYBELLA® determined after review of the subject's medical history for which the evaluating investigator identifies no clinically significant abnormality.
* Subject has read and signed the study written informed consent form.

Exclusion Criteria

* Body Mass Index ≥40 as determined at screening.
* Subject has excessive skin laxity, as determined by the evaluating investigator, in the neck or chin area or other anatomical feature (e.g., predominant subplatysmal fat, loose skin in the neck or chin area, prominent platysmal bands) for which reduction in the submental fat may result in an aesthetically unacceptable outcome.
* There is evidence of any cause of enlargement in the submental area (e.g., thyroid enlargement, cervical adenopathy) other than localized submental fat.
* Subject has a history of trauma associated with the chin or neck areas, which in the judgement of the investigator may affect evaluation of safety or efficacy of treatment.
* Subject has a history of treatment with CoolSculpting or KYBELLA® in the intended treatment area or has a history of any intervention to treat submental fat (e.g., liposuction, surgery, or lipolytic agents).
* Subject has a history of treatment with radiofrequency, micro-focused ultrasound, laser procedures, chemical peels, or dermal fillers in the neck or chin area within 12 months before the first treatment session.
* Subject has a history of treatment with botulinum toxin injections in the neck or chin area within 6 months before the first treatment session.
* Subject has a known history of cryoglobulinemia, cold urticaria, paroxysmal cold hemoglobinuria or cold agglutinin disease.
* Subject has a known history of Raynaud's disease, or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of facial nerve paresis or paralysis (such as Bell's palsy)
* Subject has a history or current symptoms of dysphagia.
* Subject has a history of prior neck surgery, or prior surgery in the area of intended treatment, or implant in or adjacent to the area of intended treatment.
* Subject has a history of sensitivity to any components of the KYBELLA® or to topical or local anesthetics (e.g., lidocaine, benzocaine, novocaine).
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is currently taking or has taken diet pills or weight control supplements within the past month.
* Subject has any dermatological conditions, such as scars in the location of the treatment area that may interfere with the treatment or evaluation.
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system.
* Women of childbearing potential not using a reliable means of contraception.
* Subject is unable or unwilling to comply with the study requirements.
* Subject has received treatment with an investigational device or agent within 30 days before the subject's first treatment session.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Jiang, NP, Study Director — Zeltiq Aesthetics
Locations (1):
- Rebecca Fitzgerald, MD Dermatology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella: All subjects enrolled in the study were to receive 2 CoolSculpting sessions in which submental fat was treated. Six weeks following the final CoolSculpting session, subjects were treated with Kybella in the submental area.
Period: Overall Study
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43 [24 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 16
  Hispanic | 0
  African American | 0
  Other | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
BMI [Mean (Full Range); unit: kg/m^2] | 31.8 [25.1 to 39]

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Have at Least a 1-grade Improvement on the Clinician Reported Submental Fat Rating Scale (CR-SMFRS) at the Final Follow-up Visit When Compared to the Baseline Grade.
Description: The CR-SMFRS is a 5-point scale ranging from 0 to 5, with '0' = Absent Submental Convexity: no localized submental fat evident, '1' = Mild Submental Convexity: minimal localized submental fat, '2'= Moderate Submental Convexity: prominent, localized submental fat, '3' = Severe Submental Convexity: Marked, localized submental fat, '4' = Extreme Submental Convexity. The investigator performed the evaluation of each subject, including palpation of the neck and chin area; oblique anterior and profile views of the chin and neck; and observation of pronation, supination and lateral movement of the head. The score was determined during a live assessment while the subject's head was in the Frankfort plane posture and was recorded as a whole number.
Time Frame: Baseline and 12-week post-treatment follow-up visit.
Population: Of the 16 subjects enrolled in the study, 1 subject withdrew after the first CoolSculpting treatment, an another subject was excluded from the efficacy analysis due to failure to maintain weight according to protocol requirements.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
Number analyzed (Participants) | 14
Participants | 14

2. Primary Outcome: The Proportion of Subjects for Whom a 2-grade Improvement Was Recorded Using the CR-SMFRS From Baseline to Final Follow-uo Visit.
Description: as for outcome 1
Time Frame: Baseline and 12-week post-treatment follow-up visit.
Population: Of the 16 subjects enrolled in the study, 1 subject withdrew from the study after the first CoolSculpting treatment. A second subject was excluded from the efficacy analysis for weight change outside of the range specified in the study protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
Number analyzed (Participants) | 14
Participants | 10

3. Primary Outcome: The Number of Device, Drug or Procedure-related Adverse Events.
Description: Adverse event information is collected from the time of study enrollment to the completion of the final follow-up visit. Investigators determined if adverse events occurring in the study are 'Not Related', 'Possibly Related', 'Probably Related', or have a 'Causal" relationship to the study device, drug or procedure.
Time Frame: 12-week post-treatment follow-up visit, approximately 31 weeks from enrollment.
Population: All adverse events for all subjects treated with CoolSculpting or CoolSculpting and Kybella were evaluated for the relationship to the device, the drug or the study procedure.
Measure: Number; unit: adverse events
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
Number analyzed (Participants) | 16
adverse events | 90

4. Secondary Outcome: Change in Submental Fat Layer Thickness as Measured by Ultrasound.
Description: Change in the fat layer thickness will be calculated by comparison of pre-treatment and 12 week post-final treatment ultrasound measurements taken in the area treated with the device. The Sponsor's standardized techniques for obtaining ultrasound imaging will be used. Overall fat layer thickness changes will be normalized for each subject by subtracting the change in the pre-treatment area from the change in treated area to remove the influence of weight variations. This result is considered the treatment effect. Results indicate the fat layer reduction in centimeters.
Time Frame: 12-week post-treatment follow-up visit.
Population: Of the 16 subjects enrolled and treated, 1 subject withdrew from the study after the first CoolSculpting treatment. A second subject was excluded from the efficacy analysis for weight gain outside of protocol requirements.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
Number analyzed (Participants) | 14
centimeters | 0.02 (0.13)

5. Secondary Outcome: Subject Satisfaction as Measured by a Comparison of Baseline and 12-weeks Post-final Treatment of Completed Subject Self-Rating Scales (SSRS).
Description: The SSRS is a 7-point scale with 0 = extremely dissatisfied 1= dissatisfied, 2 = slightly dissatisfied, 3 = neither satisfied nor dissatisfied, 4 = slightly dissatisfied, 5 = satisfied, and 6 = extremely satisfied. The percentage of subjects reporting "slightly satisfied", "satisfied" or "extremely satisfied" is presented.
Time Frame: Baseline and 12-weeks post- final treatment visit.
Population: Of the 16 subjects enrolled and treated in the study, 1 subject withdrew from the study after the first CoolSculpting treatment. Another subject was excluded from this efficacy analysis for weight gain outside requirements defined in the study protocol.
Measure: Mean (95% Confidence Interval); unit: percent of participants
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
Number analyzed (Participants) | 14
percent of participants | 71.4 [41.9 to 91.6]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time of enrollment through the final 12-week post-treatment follow-up visit. The final follow-up visit timing was predicated on the number of Kybella treatment sessions each subject completed. The range for the final follow-up visit was from 28 to 31 weeks.
Arm/Group | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 15/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment for Submental Fat Reduction Using Zeltiq CoolSculpting System Followed by Kybella (N=16)
Erythema/purpura (Skin and subcutaneous tissue disorders) | 15 (28)
Edema (Skin and subcutaneous tissue disorders) | 15 (29)
Numbness (Skin and subcutaneous tissue disorders) | 15 (25)
Numbness and tingling (Skin and subcutaneous tissue disorders) | 4 (4)
Bruising (Skin and subcutaneous tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Foot sprain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/98/NCT03510598/Prot_SAP_000.pdf